CLINICAL TRIAL: NCT07213089
Title: A Phase II/III Randomized, Observer-blind, Active-controlled Study to Compare Non-inferior Immunogenicity of a DTaPgen Vaccine to a Licensed DTaP-IPV, When Administered to Healthy Toddlers Aged of 15-36 Months Old.
Brief Title: Immunogenicity of a Combined Diphtheria-Tetanus-recombinant Acellular Pertussis (DTaP) Vaccine in Healthy Toddlers
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: BioNet-Asia Co., Ltd. (Industry)
Collaborators: National Science and Technology Development Agency, Thailand (Other Government); Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DTA201; TCTR20200325002 (Registry Identifier: Thai Clinical Trials Registry)
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Pertussis Whooping Cough
Keywords: Pertussis Whooping cough
MeSH Terms: interventions — Vaccines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combined Diphtheria-Tetanus-recombinant acellular pertussis (DTaP) vaccine (Experimental): Participants who having completed the 3 doses DTwP or 3-dose DTaP vaccination (on interchange of DTwP and DTaP during primary immunization) will be randomized to receive Acellular pertussis (DTaP) vaccine (0.5 ml) given by intramuscularly as a single dose
  Interventions: Biological: Combined Diphtheria-Tetanus-recombinant acellular pertussis (DTaP) vaccine
- Licensed DTaP (Active Comparator): Participants who having completed the 3 doses DTwP or 3-dose DTaP vaccination (on interchange of DTwP and DTaP during primary immunization) will be randomized to receive Acellular pertussis (DTaP) vaccine (0.5 ml) given by intramuscularly as a single dose
  Interventions: Biological: Licensed DTaP

INTERVENTIONS:
Biological: Combined Diphtheria-Tetanus-recombinant acellular pertussis (DTaP) vaccine — A single dose of Acellular pertussis (DTaP) vaccine 0.5 ml will be given by intramuscularly at Day 0
  Arms: Combined Diphtheria-Tetanus-recombinant acellular pertussis (DTaP) vaccine
Biological: Licensed DTaP — A single dose of Acellular pertussis (DTaP) vaccine 0.5 ml. will be given by intramuscular as at Day 0
  Arms: Licensed DTaP

SUMMARY:
Recombinant acellular pertussis vaccines containing genetically detoxified Pertussis Toxin (PTgen) have been used for booster immunisation in children, adolescents and adults including pregnant women in Thailand. Three vaccines have been licensed in Thailand, a monovalent (aPgen) and two vaccines combined with tetanus and reduced diphtheria dose vaccines (TdaPgen and Tdapgen). To address the need for improved vaccines in younger children, a new recombinant pediatric DTaP vaccine (DTaPgen) containing 5 µg genetically detoxified Pertussis Toxin (PTgen) and 10 µg Filamentous Hemagglutinin (FHA) was developed and found safe and immunogenic in a phase II trial in children aged 3 years onwards.

The purpose of this study is to assess the immunogenicity and safety of this new pediatric formulation DTaPgen given as the first booster dose in healthy toddlers aged 15 to 36 months compared to a commercially available vaccine in Thailand.

DETAILED DESCRIPTION:
This is a phase II/III randomized, observer-blind, active-controlled study conducted in Thailand, children aged 15-36-month-old with a history of DTwP (n=240) or DTaP (n=50) priming were randomized 2:1 to receive a dose of recombinant DTaPgen or licensed DTaP-IPV. The aim of this study is to evaluate the safety and non-inferior immunogenicity of DTaPgen versus DTaP-IPV vaccine given as the first booster dose in toddlers.

Safety up to 1-year and vaccine antibody persistence will also be assessed for all children.

ELIGIBILITY:
Inclusion Criteria: Participants will be eligible for inclusion if ALL of the following criteria are met at the time of screening:

1. 15 to 36 months of age at the time of vaccination.
2. Having completed the 3-dose DTwP or 3-dose DTaP vaccination (no interchange of DTwP and DTaP during primary immunization).
3. The parents or legal guardians of the participant are able to read and write.
4. The parents or legal guardians can provide written informed consent.
5. Healthy, as established by pertinent medical history and physical examination.

Exclusion Criteria: A participant with ANY of the following criteria at study entry will not be eligible for participation

1. History of any significant medical illness such as, but not limited to, immune deficiency, renal, hepatic, cardiovascular, or endocrine disorder as determined by the investigator based on medical history and physical examination.
2. History of allergy or hypersensitivity to any vaccine (including its component).
3. History of any serious adverse event or neurological adverse event after vaccination.
4. Having received only 1 or 2 doses of DTwP or DTaP (incomplete primary immunization) after birth until the study enrollment.
5. Having received the 4th dose DTwP or DTaP vaccination.
6. Having experienced a physician diagnosed diphtheria or tetanus or pertussis illness within 1 year prior to recruitment.
7. Receipt of any vaccine within 28 days prior to enrollment (3 months for live-attenuated vaccines).
8. Planning to receive tetanus, diphtheria, pertussis or planning to participate in another clinical trial during the study period (approximately 1 year).
9. Receipt of blood or blood component or immunoglobulin within 3 months prior to recruitment.
10. History of receiving any immunosuppressive drug or systemic corticosteroid (more than 0.5 mg/kg of prednisolone or equivalent for more than 14 days) within 3 months prior to recruitment.
11. Any bleeding disorder.
12. Any abnormality of splenic or thymic function.
13. Any progressive or severe neurological disorder such as seizure disorder or Guillain- Barre syndrome;
14. History of any illness including cognitive impairment and psychiatric disease that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the participants due to participation in the study.
15. Fever as defined by body temperature more than 38 degree celsius at the time of enrollment (temporary exclusion criterion).

Ages: 15 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 290 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-05-12 (Actual)

PRIMARY OUTCOMES:
Seroconversion rates of PT | At 28 days following vaccination
  ELISA

SECONDARY OUTCOMES:
Percentages of participants with solicited post-immunization local and systemic reactions | During 7 days following vaccination
  Self assessment by participant and data record from Diary Card
Percentages of participants with AEs | During 28 days following vaccination
  AEs reported by participant
Percentages of participants with SAEs | During 28 days following vaccination
  SAEs reported by participant
GMT antibody concentration to anti-PT neutralizing antibody | Baseline and Day 28 after vaccination
  CHO
GMT antibody concentration to DT, TT, PT and FHA | Baseline and Day 28 after vaccination
  ELISA
Seroprotection rates of Tetanus and Diphtheria | Day 28 after vaccination
  ELISA
Seroconversion rates of FHA and anti-PT neutralizing antibody | Day 28 after vaccination
  ELISA and CHO
Percentages of participants with SAEs | Day 336 after vaccination
  SAEs reported by participant
Seroconversion rates of FHA and anti-PT neutralizing antibody | Day 336 after vaccination
  ELISA and CHO
GMT antibody concentration to DT, TT, PT and FHA | Day 336 after vaccination
  ELISA
GMT antibody concentration to anti-PT neutralizing antibody | Day 336 after vaccination
  CHO
Seroprotection rates of Tetanus and Diphtheria | Day 336 after vaccination
  ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Punnee Pitisuttithum, Principal Investigator — Vaccine Trial Centre (VTC), Faculty of Tropical Medicine, Mahidol University
Locations (3):
- Thailand (3):
  - Vaccine Trial Centre (VTC), Faculty of Tropical Medicine, Mahidol University, Bangkok, Bangkok
  - Kamphaengphet Hospital, Kamphaeng Phet, Changwat Kamphaeng Phet
  - Phaholpolpayuhasena Hospital, Kanchanaburi, Kanchanaburi

IPD SHARING:
Plan to Share IPD: No
Undecided